CLINICAL TRIAL: NCT01775098
Title: Allopurinol in Acute Gout The Title Will Not be Change as the Study as Been Closed.
Brief Title: Allopurinol in Acute Gout
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: because of a lack of funding
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Artur de Brum-Fernandes, Doctor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Allopurinol in acute gout
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Gout
Keywords: Gout; uric acid; allopurinol
MeSH Terms: conditions — Gout | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allopurinol (Experimental): treatment with allopurinol
  Interventions: Drug: allopurinol
- placebo (Placebo Comparator): placebo comparator
  Interventions: Drug: allopurinol

INTERVENTIONS:
Drug: allopurinol — No arms will not be change as the study as been closed.

SUMMARY:
The objectives of the present study are to determine if starting treatement of hyperuricemia with allopurinol during an acute gout crises has an impact on the duration or the severity of the crises

ELIGIBILITY:
Inclusion Criteria:

More than 18 years old Able to sign informed consent Indication of long-term treatment with allopurinol Acute gout crisis

Exclusion Criteria:

Les than 18 years-old Unable to consent Contra-indication to allopurinol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Duration of the gout crises | First 7 days after visit
  Presence of inflammatory signs